CLINICAL TRIAL: NCT01377181
Title: Phase 3 Study of Laparoscopic Hernia Repair With Lateral Umbilicus Ligament for Children
Brief Title: Laparoscopic Hernia Repair With Lateral Umbilicus Ligament for Children
Status: Completed | Type: Observational
Sponsor: The Second People's Hospital of GuangDong Province (Other)
Responsible Party: Kaiyun Chen, The Second People's Hospital of GuangDong Province
Other Study IDs: ABT-1233-RV
Record Dates: First submitted 2010-09-02; First posted 2011-06-21 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2000-01

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Laparoscope; Lateral us ligament; Recurrence; Pediatric; unilateral inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group A: the patients were accepted laparoscopic purse-string knot closing the internal hernia opening only
- group B: the patients were accepted the lateral umbilicus ligament covering the internal hernia opening region after the laparoscopic purse-string knot

SUMMARY:
The role of laparoscopic surgery in pediatric inguinal hernia repair is clear. Laparoscopic hernia repair is especially advantageous for bilateral diseases and minimally invasive technique in children because it avoids vas injury. However, the problem of recurrent rate has not been resolved. The aim of this study was to refine the current criteria used the lateral umbilicus ligament covering the internal hernia opening region, and eliminated recurrence in laparoscopic inguinal hernia (LIH) repair in children. The investigators hypothesized that the lateral umbilicus ligament covering the internal hernia opening region after the laparoscopic purse-string knot would result in lower recurrence and the same operation relative complication

DETAILED DESCRIPTION:
The primary outcome measure was the recurrence rate after surgery, and the secondary outcome measures included degree of postoperative pain, the amount of postoperative analgesia, procedural duration, number of days to recovery normal activity, surgical complications, cosmetic results, and patient satisfaction. The outcome was recorded at the outpatient visits 10 days, 6 months, 1 year, 3 years and 5 years after the surgery. The cosmetic result was scored (unsatisfactory = 0, satisfactory = 1, good = 2, and excellent = 3) by the patients or parents, the attending nurse, and the surgeon (maximum points = 9). The patient satisfaction was scored similarly (unsatisfactory = 0, satisfactory = 1, good = 2, and excellent = 3). The long axis of the testes was measured.

ELIGIBILITY:
Inclusion Criteria:

* unilateral inguinal hernia
* age between 2 years and 17 years
* no history of abdominal or inguinal operations
* the age range was based on the day surgery criteria of our hospital
* of male patients, only those with completely descended testes were included

Exclusion Criteria:

* the bilateral hernia
* the recurrence hernia

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All patients between 2 years and 17 years of age undergoing laparoscopic inguinal hernia repair at our institution by a single surgeon from January, 2000 to August, 2005 were prospectively followed for outcome.
Sampling Method: Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2000-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
recurrence rate | five years
  the inguinal hernia recurrence after operation

SECONDARY OUTCOMES:
number of days to recovery normal activity | one month
  the days to recovery normal activity after surgery
degree of postoperative pain | one year
  postoperative pain was recorded on a modified objective pain scale (OPS) from 0 to 9.9. The next morning following discharge, a nurse specialist blinded to the operative approach phoned the families and recorded the level of pain on a scale from 0 to 3 (no pain = 0, mild pain = 1, moderate pain = 2, severe pain = 3)

CONTACTS AND LOCATIONS:
Overall Officials: kaiyun chen, MD, Study Chair — The Second People's Hospital of GuangDong Province
Locations (1):
- The Second People's Hospital of GuangDong Province, Guangzhou, Guangdong, China